CLINICAL TRIAL: NCT04833933
Title: Impact of Primary Care COPD Screening Strategies on the Smoking Cessation Process at 2 Years Follow-up of the Randomized, Multicenter, Clustered Controlled Trial DISCO
Brief Title: Impact of Primary Care COPD Screening Strategies on the Smoking Cessation Process (DISCO-SET)
Acronym: DISCO-SET
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC21_9742_DISCO-SET
Record Dates: First submitted 2021-04-02; First posted 2021-04-06 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Smoking Cessation; Pulmonary Disease, Chronic Obstructive
Keywords: Tobacco use cessation devices; Electronic Nicotine Delivery Systems; Cross-Sectional Studies; Smokers; Primary Care
MeSH Terms: conditions — Smoking Cessation; Pulmonary Disease, Chronic Obstructive; Vaping

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Control group: Initially in DISCO trial : no intervention, usual care
  In DISCO-SET trial : survey (the same in the 4 groups)
  Interventions: Other: Phone survey about smoking cessation process since intervention in DISCO trial
- Questionnaire: Initially in DISCO trial : Targeted screening of COPD by GPs via the GOLD / HAS questionnaire. The questionnaire includes 4 questions for patients over 40. At least one positive response is an indication to perform a spirometry.
  In DISCO-SET trial : survey (the same in the 4 groups)
  Interventions: Other: Phone survey about smoking cessation process since intervention in DISCO trial
- Coordination: Initially in DISCO trial : Information of the GPs of the existence of a coordination of the care of proximity to facilitate the access to the spirometry (identification of a referent specialist, making appointments).
  In DISCO-SET trial : survey (the same in the 4 groups)
  Interventions: Other: Phone survey about smoking cessation process since intervention in DISCO trial
- Questionnaire + Coordination: Initially in DISCO trial :
  * Targeted screening of COPD by GPs via the GOLD / HAS questionnaire. The questionnaire includes 4 questions for patients over 40. At least one positive response is an indication to perform a spirometry.
  * Information of the GPs of the existence of a coordination of the care of proximity to facilitate the access to the spirometry (identification of a referent specialist, making appointments).
  In DISCO-SET trial : survey (the same in the 4 groups)
  Interventions: Other: Phone survey about smoking cessation process since intervention in DISCO trial

INTERVENTIONS:
Other: Phone survey about smoking cessation process since intervention in DISCO trial — We will conduct a phone survey at 2 years follow-up with a random sample of smoking patients at inclusion in DISCO trial, to know the evolution of their smoking habits, the quit attempts since the intervention and the modalities of these attempts.

SUMMARY:
The general practitioner is confronted with unselected smokers whose attempts to quit smoking are often repeated over time before leading to a definitive cessation.

Each year, 3-5% of smokers succeed in quitting in the general population. The corollary is that the majority of smokers are in a situation of failure in their attempt to quit: 33% declared during the 2019 French Health Barometer to have made an attempt of at least 7 days in the past year. Thus, this status of "smoker" can cover a wide variety of situations: no attempt to stop smoking, attempt(s) of more or less clinical significance, previous support or not by a health professional, etc. Currently, the HAS recommendations do not determine a specific course of action for these smokers, whose experiences may be very different. It could therefore be interesting to objectivize the smoking cessation process of these patients who have or have not succeeded in quitting, in order to deduce profiles of smokers according to their previous smoking cessation experiences. Furthermore, the choice and relevance of the cessation criteria used are debated.

Following the randomized controlled trial DISCO on COPD screening interventions in primary care (3 intervention arms, 1 control arm), the investigators will carry out a pilot cross-sectional survey on the cessation process of smokers during the 2 years following their participation, evaluating the incidence and modalities of cessation attempts of smokers belonging to an age group at risk of COPD (40-80 years) and who initially consulted their general practitioner for any reason 2 years ago at the time of their inclusion.

The impact on future management could be the personalization of cessation advice given to smokers according to quantitative and qualitative indicators specific to their experience, their previous history of smoking cessation, their health situation and socio-demographic characteristics. Eventually, a gradation of the levels of support offered to patients in general practice on the basis of predictive factors of smoking cessation could be studied.

The investigators hypothesize that participation in COPD screening with the GP may be associated with patient progress in quitting smoking. This pilot study will be conducted on a random sample of 120 participants from the subgroup of 544 patients who were smokers at inclusion in DISCO.

ELIGIBILITY:
Inclusion Criteria:

* Active smoker patient at inclusion in the DISCO study,
* No objection to participate in the study,
* Patient still followed in the active file of general practitioners' offices (GP).
* Patient's telephone and postal details available

Exclusion Criteria:

* Patient not physically or mentally able to complete the phone survey,
* Patient deceased,
* Patient not reachable despite 5 phone calls and message left on answering machine.
* Patient under curatorship, guardianship or safeguard of justice

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Random sample of 120 patients from the subgroup of 544 patients who were active smokers at inclusion in the DISCO study two years ago
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-04-07 (Actual); Primary Completion 2021-07-07 (Actual); Study Completion 2021-07-07 (Actual)

PRIMARY OUTCOMES:
Percentage of smoking patients with at least 1 episode of smoking cessation attempts of at least 28 days since inclusion in the DISCO study. | 2 years

SECONDARY OUTCOMES:
Smoking cessation of at least 7 days | 2 years
  Number of patients with smoking cessation of at least 7 days in patients who had quit smoking by the day of the survey, since inclusion in DISCO study
Smoking cessation of at least 28 days | 2 years
  Number of patients with smoking cessation of at least 28 days in patients who had quit smoking by the day of the survey, since inclusion in DISCO study
Smoking cessation of at least 6 months | 2 years
  Number of patients with smoking cessation of at least 6 months in patients who had quit smoking by the day of the survey, since inclusion in DISCO study
Smoking cessation attempts of 7 days | 2 years
  Number of patients with smoking cessation attempts of 7 days in active smoking patients at the day of the survey, since inclusion in DISCO
Smoking cessation attempts of 28 days | 2 years
  Number of patients with smoking cessation attempts of 28 days in active smoking patients at the day of the survey, since inclusion in DISCO
Smoking cessation attempts of 6 months | 2 years
  Number of patients with smoking cessation attempts of 6 months in active smoking patients at the day of the survey, since inclusion in DISCO
Cumulative duration (days) of smoking cessation attempts since inclusion in DISCO study | 2 years
Change in daily tobacco consumption in cigarettes per day, compared to the consumption reported at inclusion in DISCO | 2 years
Change in daily tobacco consumption in cigarettes per day at least 50% on the day of the survey, compared to the consumption reported at inclusion in DISCO | 2 years
Percentage of patients who made their first smoking cessation attempt in their life since their inclusion in the DISCO study | 2 years
Percentage of patients who used each kind of heath professionnal aid and material cessation aid since their inclusion in the DISCO study | 2 years
Percentage of patients who have discussed smoking with their general practitioner and number of consultations where this was discussed since their inclusion in the DISCO study | 2 years
Percentage of general practitioners still in practice, available for this study and who have not changed their patient base | 2 years
Percentage of patients included with completed questionnaires in the sample of 120 patients, with percentage of refusals to participate, incomplete questionnaires and non-responders | 2 years
Average number of calls per patient before inclusion and per patient included with completed questionnaire | 2 years
Average number of trips per practitioners and per number of patients included in each practitioners | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bruno LAVIOLLE, PhD, Study Chair — Rennes UH; Anthony CHAPRON, PhD, Principal Investigator — Faculty of medicine of rennes; Anthony CHAPRON, PhD, Study Director — Faculty of medicine of rennes
Locations (12):
- France (12):
  - Emmanuelle FOURE-AMELOT, Bédée, Brittany Region
  - Béatrice NEGARET, Breteil, Brittany Region
  - Lucie DELATTE, Janzé, Brittany Region
  - Marie BROSSET, Miniac-Morvan, Brittany Region
  - Antoine MOUTEL, Redon, Brittany Region
  - Anna JARNO-JOSSE, Rennes, Brittany Region
  - Hoël CHARBONNEL, Rennes, Brittany Region
  - Romain NIFENECKER, Rennes, Brittany Region
  - Jean-Philippe DUGUEY, St-Malo, Brittany Region
  - Laurent LENOBLE, Sulniac, Brittany Region
  - Lucie MURGALE, Talensac, Brittany Region
  - Marieke SALACROUP, Tremblay, Brittany Region

IPD SHARING:
Plan to Share IPD: Undecided